CLINICAL TRIAL: NCT04921475
Title: Association of Renal Regional Oxygen Saturation and Postprocedural Acute Kidney Injury in Patients Undergoing Transcatheter Aortic Valve Implantation
Brief Title: Renal Regional Oxygen Saturation During Transcatheter Aortic Valve Implantation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, PhD, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: TAVI_renalRSO2
Record Dates: First submitted 2021-06-07; First posted 2021-06-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Kidney Injury, Acute; Transcatheter Aortic Valve Implantation
Keywords: renal regional oxygen saturation; acute kidney injury; transcatheter aortic valve implantation
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal regional oxygen saturation: Renal regional oxygen saturation is measured by using near infrared spectroscopy during transcatheter aortic valve implantation
  Interventions: Device: Regional oxygen saturation monitoring

INTERVENTIONS:
Device: Regional oxygen saturation monitoring — Regional oxygen saturation of kidney is monitored using near infrared spectroscopy

SUMMARY:
This prospective observational study evaluates the association of peri-procedural changes in renal regional oxygen saturation and post-procedural acute kidney injury in patients undergoing transcatheter aortic valve implantation.

DETAILED DESCRIPTION:
This prospective observational cohort study evaluated the association of renal regional oxygen saturation, measured during transcatheter aortic valve implantation, and post-procedural acute kidney injury. Renal regional oxygen saturation is measured using near-infrared spectroscopy on the skin surface over the kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 20 years old) undergoing transcatheter (transfemoral) aortic valve implantation

Exclusion Criteria:

* Emergent procedure
* Pre-procedural severe renal impairment (eGFR < 30 mL/min/1.73 m2)
* Pre-procedural hemodialysis
* Distance from skin to renal capsule > 4 cm
* Pre-procedural mechanical ventilation
* Refuse to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age >= 20 years) undergoing transfemoral transcatheter aortic valve implantation are eligible for this observational study.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | during 7 days post-TAVI
  increase in serum creatinine compared with baseline or reduced urine output

SECONDARY OUTCOMES:
composite complication | during 7 days post-TAVI or until discharge
  stroke, delirium, acute MI, heart failure, new or worsening arrhythmia, mechanical ventilation over 24 h, length of ICU stay, hospital stay, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee HS, Cho YJ, Yoo S, Lee S, Ju JW, Nam K, Jeon Y. Association of renal regional tissue oxygen saturation and post-procedural acute kidney injury following transcatheter aortic valve implantation. J Clin Monit Comput. 2025 Dec;39(6):1203-1213. doi: 10.1007/s10877-025-01339-2. Epub 2025 Aug 13. PMID 40802215